CLINICAL TRIAL: NCT04105413
Title: Early Diagnosis of Neonatal Sepsis Using Modified Hematological Scoring System
Brief Title: Early Diagnosis of Neonatal Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fady Magdy Saber, principle investigator, Assiut University
Other Study IDs: EDONS
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Sepses, Neonatal
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood culturs — CBC, Blood culture and CRP

SUMMARY:
Sepsis is defined as a systemic inflammatory response syndrome (SIRS) associated with infection diagnosed either on microbiologic cultures or strong clinical evidence of an infection.

DETAILED DESCRIPTION:
Sepsis is defined as a systemic inflammatory response syndrome (SIRS) associated with infection diagnosed either on microbiologic cultures or strong clinical evidence of an infection..Worldwide, neonatal sepsis is responsible for 4 million deaths annually and 99% of them occur in developing countries.. . morbidity associated with sepsis includes sensorineural hearing loss, visual disturbances, seizures, and neurodevelopmental issues.. Blood culture is considered as gold standard for diagnosis of sepsis. The ideal diagnostic test should be inexpensive, have quick results Hematologic scoring system(HSS) of Rodwell et al. includes the following: a) White blood cell and platelet count b) White blood differential count c) Nucleated red blood cell count (to correct WBC count) d) Assessment of neutrophil morphology for degenerative changes. A modified HSS(modified hematological scoring system) was developed by removing the repetitive parameters, adding a new parameter - nucleated RBC.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with history of prolonged rupture of membranes, maternal intrapartum fever or non specific signs of sepsis namely; neonatal fever or hypothermia , poor feeding ,lethargy, irritability, depressed neonatal reflexes ,respiratory distress including apnea or cyanosis,hypoxia,poor capillary perfusion,bradycardia,hypotension,pallor,edema,vomiting,diarrhea,abdominal distention, bulging anterior fontanelle,coma,seizures,unexplained jaundice, reduced suckling, bleeding problems,hypoglycemia,hyperglycemia or metabolic acidosis were included in the study

Exclusion Criteria:

* All the newborn babies with history of delayed cry, meconium aspiration, congenital anomaly, history of antibiotics administration prior to admission to the baby or mother, intrapartum and neonatal death in sibling with similar presentation will be excluded

Max Age: 28 Days | Sex: All
Age Groups: Child
Study Population: all neonates suspected neonatal sepsis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-30 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Early detection of neonatal sepsia | average 1 year
  To determine the accuracy of a simple and cost effective Modified hematological scoring system in the early diagnosis of neonatal sepsis using blood culture as a gold standard in neonates attending Neonatology Unit of Assiut University Children Hospital

REFERENCES:
- [Background] Wynn J, Cornell TT, Wong HR, Shanley TP, Wheeler DS. The host response to sepsis and developmental impact. Pediatrics. 2010 May;125(5):1031-41. doi: 10.1542/peds.2009-3301. Epub 2010 Apr 26. PMID 20421258
- [Background] Darmstadt GL, Saha SK, Choi Y, El Arifeen S, Ahmed NU, Bari S, Rahman SM, Mannan I, Crook D, Fatima K, Winch PJ, Seraji HR, Begum N, Rahman R, Islam M, Rahman A, Black RE, Santosham M, Sacks E, Baqui AH; Bangladesh Projahnmo-2 (Mirzapur) Study Group. Population-based incidence and etiology of community-acquired neonatal bacteremia in Mirzapur, Bangladesh: an observational study. J Infect Dis. 2009 Sep 15;200(6):906-15. doi: 10.1086/605473. PMID 19671016
- [Background] Mishra UK, Jacobs SE, Doyle LW, Garland SM. Newer approaches to the diagnosis of early onset neonatal sepsis. Arch Dis Child Fetal Neonatal Ed. 2006 May;91(3):F208-12. doi: 10.1136/adc.2004.064188. PMID 16632649
- [Background] Rodwell RL, Leslie AL, Tudehope DI. Early diagnosis of neonatal sepsis using a hematologic scoring system. J Pediatr. 1988 May;112(5):761-7. doi: 10.1016/s0022-3476(88)80699-1. PMID 3361389
- [Background] Mikhael M, Brown LS, Rosenfeld CR. Serial neutrophil values facilitate predicting the absence of neonatal early-onset sepsis. J Pediatr. 2014 Mar;164(3):522-8.e1-3. doi: 10.1016/j.jpeds.2013.10.080. Epub 2013 Dec 10. PMID 24331688